CLINICAL TRIAL: NCT05843786
Title: Human Recombinant Interferon Gamma in the Treatment of Ventilator-acquired Pneumonia in ICU Patients
Acronym: IGNORANT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL22_0851; 2022-502229-16-00 (Other: EUCT number)
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Critical Illness; Interferon-gamma; Immunodepression; Sepsis; Trauma; Monocyte HLA-DR; immunostimulation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Critical Illness; Sepsis; Wounds and Injuries | interventions — Interferon-gamma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferon gamma treatment (Experimental): Interferon gamma treatment (100 micrograms /day during 5 days)
  Interventions: Drug: Interferon gamma
- Placebo (Placebo Comparator): The comparator drug (placebo) is an injectable solution of sodium chloride 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon gamma — Daily subcutaneous administration of Interferon gamma during 5 days
  Arms: Interferon gamma treatment
Drug: Placebo — Placebo during 5 days
  Arms: Placebo

SUMMARY:
Clinical presentation of patients after severe injury such as a severe infection, trauma or extensive burns is characterized by the simultaneous occurrence of dysregulation of the initial inflammatory response and immunosuppression associating quantitative and functional alterations of innate and adaptive immune cells. These acquired immune dysfunctions have been associated with an increased susceptibility to nosocomial infections, foremost among which are ventilator-associated pneumonia (VAP). Despite the implementation of a set of preventive measures, the incidence of these VAP remains high in intensive care, with rates in Europe of 1.5% per day of ventilation.

Post-aggressive immunosuppression is characterized by the decrease in the expression of HLA-DR (belonging to the type II major histocompatibility complex, MHC-II) on the surface of monocytes (mHLA-DR). The administration of interferon gamma (IFNγ) can restore the level of mHLA-DR and may possibly improve the prognosis as an adjuvant therapy associated to antibiotics. However, the level of proof of this therapeutic strategy is low, limited to small cohorts of patients, or clinical studies without prior immunodepression assessment. The objective of this study is to conduct a randomized, double-blind, placebo-controlled superiority trial to assess the effect of IFNγ administration on the duration of mechanical ventilation following the first episode of VAP in patients having an HLA-DR < 8000 AB/C

All reported data about recombinant human IFNγ 1b for the control of secondary infections in patients with septic shock used the dose of 100 micrograms per day by subcutaneous route for 3 to 5 days . At this dose, no retrospective study has reported any serious adverse effects and recombinant human IFNγ 1b allows an increase in monocyte membrane expression of mHLA-DR.

ELIGIBILITY:
Inclusion Criteria:

* adult patients hospitalized in intensive care unit
* under mechanical ventilation for more than 5 days
* having a first episode of VAP (with a Clinical Pulmonary Infectious Score (CPIS score) >6)
* treated with antibiotics for less than 24 hours
* with monocyte HLA-DR < 8000 AB/C
* written informed consent signed by the patient's trusted support person, or in the absence of the patient's representative and taking into account the agreement of the relative obtained by telephone emergency certificate completed and signed by the investigator
* membership of a social security scheme

Exclusion Criteria:

* inability to administer the first dose of treatment in the study within 48 hours of the start of antibiotic therapy (antibiotic therapy for VAP)
* Noradrenaline > 0.25 mcg/kg/min
* Immunosuppression, defined by:

  * solid tumor with chemotherapy in the last 3 months
  * progressive metastatic disease
  * hematological disease
  * solid organ transplantation
  * HIV infection (AIDS stage or not)
  * corticosteroid therapy at any dose for more than 3 months
  * ≥ 1 mg/kg of Prednisone equivalent for more than 7 days
  * immunosuppressive therapy
* Head and/or cervical spine trauma : with a predictable impact on the duration of mechanical ventilation (left to the investigator's judgement), the investigator will assess whether the patient meets the following neurological criteria for extubation during their recovery:
* A level of consciousness assessed as 0 or 1 on the Richmond Agitation-Sedation Scale (RASS)
* FiO2 <40%
* PEEP level <5 cmH2O
* A FR/Vt ratio <105
* Effective cough
* Response to simple commands
* Administration of noradrenaline < 0.2 mcg/kg/min
* Cardiocirculatory arrest
* Burn patient
* Cirrhosis with Child B or C score
* Infection with Aspergillus spp.
* Refusal to participate
* Patient participating in another interventional research in progress or including an exclusion period still in progress at pre-inclusion (excluding interventional research of 2° not interfering with the endpoints of the study according to the judgment of the principal investigator)
* Lack of social coverage
* Patient under curatorship or guardianship
* Pregnant or breastfeeding women
* Patient admitted to intensive care for SARS-Cov2 pneumonia
* Known allergy to latex
* Hypersensitivity to the active substance (interferon gamma-1b) or known hypersensitivity to related products, such as another interferon, or to any of the following excipients: Mannitol, Disodium succinate hexahydrate, Succinic acid, polysorbate 20
* Existence of chronic heart disease with FeVG<45%
* Major hepatic impairment (total bilirubin>60 mg/L or 102 mcmol/L, equivalent to 3 SOFA points)
* thrombocytopenia <50000/mm3 (equivalent to 3 SOFA points) AST and/or ALT > 5N Lipase > 3N Severe chronic renal failure (creatinine clearance MDRD< 10 ml/min/1.73m2)
* Thrombocytopenia <50,000/mm3 (equivalent to 3 SOFA points)
* Respiratory failure requiring home oxygen therapy
* Persons under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
duration of mechanical ventilation assessed from the first day of VAP diagnosis | Day 28
  mechanical ventilation-free days (VFD) from extubation through D28. A beneficial effect of using recombinant human interferon gamma-1b would be a statistically significant increase in VFD in patients receiving study drug in this setting compared to the group receiving placebo.

SECONDARY OUTCOMES:
All-cause mortality in intensive care | Day 28
Previous positive microbiological sample at inclusion becomes negative | Day 5
  Previous positive microbiological sample at inclusion becomes negative, i.e. pulmonary, urinary, blood cultures
Length of stay in intensive care unit | Day 28
length of stay at hospital | Day 28
occurrence of another episode of VAP before extubation | Day 28
occurrence of another episode of infection acquired in intensive care unit | Day 28
increase of monocytic HLA-DR expression above 8000 AB/C the day after the last dose of treatment (J5) | Day 28
increase or decrease of blood leucocyte count at the day after the last dose of treatment (J5) in comparison to baseline | Day 28
Evaluation of the economic efficiency of the administration of IFN-γ (assessed by the ACER (average cost-effectiveness ratio) method) | Day 28
  Evaluation of the cost-effectiveness of IFN-γ administration (assessed by the ACER (average cost-effectiveness ratio) method)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire LUKASZEWICZ, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (9):
- France (9):
  - CHU Limoges, Limoges
  - Service civilo-militaire d'Anesthésie-Réanimation et Médecine Périopératoire, Lyon
  - Service de reanimation chirurgicale Hopital Croix-Rousse, Lyon
  - Service de reanimation médicale hôpital de la Croix-Rousse, Lyon
  - Hôpital Edouard Herriot - Médecine intensive - réanimation, Lyon
  - Service d'anesthésie-réanimation, unité de réanimation chirurgicale Picard, Nancy
  - Médecine intensive- Réanimation, Paris
  - Service d'Anesthésie-réanimation-médecine intensive Hôpital Lyon Sud, Pierre-Bénite
  - Département Anesthésie-Réanimation, Saint-Etienne